CLINICAL TRIAL: NCT06141629
Title: Benefits of a Bolus Calculator on pre-and Postprandial Glycaemic Control and Meal Flexibility of Pediatric Patients on Multiple Daily Insulin Injections
Brief Title: Benefits of a Bolus Calculator in Pediatric Patients on Multiple Daily Insulin Injections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: University of Copenhagen (Other); Hospital Sant Joan de Deu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KC19092011
Record Dates: First submitted 2023-01-26; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2011-09

CONDITIONS: Poor Glycemic Control; Quality of Life
Keywords: Metabolic control; Quality of life

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Accu-Chek Aviva Expert. (Active Comparator): Accu-Chek Aviva Expert. This is a glucometer with boluscalculator.
  Interventions: Device: accu chek Aviva Expert; Device: Accu Chek Aviva Nano
- Accu check Nano (Placebo Comparator): Accu check Nano
  Interventions: Device: accu chek Aviva Expert; Device: Accu Chek Aviva Nano

INTERVENTIONS:
Device: accu chek Aviva Expert — This bolus calculator estimates the dose of insulin to be administrated on the basis of the following parameters: current blood glucose, grams of carbohydrate, carbohydrate to insulin ratio, insulin sensitivity, target blood glucose and quantity of insulin previously administered.
Device: Accu Chek Aviva Nano — This meter is a normal glucometer without bolus calculator.

SUMMARY:
It it hypothesized that children and adolescents with type 1 diabetes, who are counting carbohydrates can achieve better metabolic control by concurrent use of the Accu-Chek Aviva Expert. Additionally, it is proposed that carbohydrate counting in combination with the the Accu-Chek Aviva Expert will lead to better quality of life as a result of fewer restrictions when eating and less variation in blood glucose.

DETAILED DESCRIPTION:
Carbohydrate (Carb) counting is a meal planning approach for patients with diabetes mellitus that focuses on carbohydrate as the primary nutrient affecting postprandial glycaemic response. In the early 1990's the Diabetes Control and Complications Trial (DCCT) used Carb counting as one of its education tools. More recently, short acting insulin analogues and insulin pumps have made the role of Carb counting important and popular. Carb counting can be used to estimate carbohydrate intake and adjust insulin around mixed meals and snacks using insulin to carbohydrate ratio. This effectively addresses the variable eating habits of most children and adolescents. Carb counting can make food planning more flexible and thus more acceptable for young patients with diabetes.

Roche has recently launched the Accu-Chek Aviva Expert recently preliminary tested in adults4, being a blood glucose meter with integrated bolus calculator and memory function. This bolus calculator estimates the dose of insulin to be administrated on the basis of the following parameters: Current blood glucose, grams of carbohydrate, carbohydrate to insulin ratio, insulin sensitivity, target blood glucose and insulin action time.

Hypothesis:

It is hypothesized that paediatric patients in MDI therapy with suboptimal regulated diabetes will achieve better glycemic control by using Accu-Chek Aviva Expert rather than carbohydrate counting alone without the use of an external calculator.

ELIGIBILITY:
Inclusion Criteria:

* - Patients with type 1 diabetes (n=120) Age > 1 year and < 18 years
* Diabetes duration >12 months
* MDI therapy (fast acting analog for meals; long acting analog as basal)
* HbA1c > 7.0% and <11%

Exclusion Criteria:

* Insulin pump therapy
* Missing consent declaration

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
better metabolic control as assessed by HbA1C | 12 months
  We hypothesize that children and adolescents with type 1 diabetes, who are counting carbohydrates can achieve better metabolic control as assessed by HbA1C.

SECONDARY OUTCOMES:
better quality of life as assessed by Hvidore questionnaire | 12 months
  quality of life as assessed by Hvidore questionnaire
better metabolic control as assessed by glucose variability | 12 months
  We hypothesize that children and adolescents with type 1 diabetes, who are counting carbohydrates can achieve better metabolic control as assessed by glucose variability by concurrent use of the Accu-Chek Aviva Expert. Additionally, we propose that carbohydrate counting in combination with the the Accu-Chek Aviva Expert will lead to better quality of life as a result of fewer restrictions when eating and less variation in blood glucose.

CONTACTS AND LOCATIONS:
Locations (1):
- UZLeuven, Leuven, Belgium